CLINICAL TRIAL: NCT00303017
Title: Safety, Efficacy and Acceptability of Flavocoxid (Limbrel) Compared With Naproxen in Subjects With Osteoarthritis of the Knee. A Pilot Study
Brief Title: Safety, Efficacy and Acceptability of Flavocoxid (Limbrel)A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Primus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Primus Protocol #OAPS
Record Dates: First submitted 2006-03-13; First posted 2006-03-15 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2008-11

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — flavocoxid; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- flavocoxid (Experimental): medical food
  Interventions: Dietary Supplement: flavocoxid
- naproxen (Active Comparator): NSAID
  Interventions: Drug: Naproxen

INTERVENTIONS:
Dietary Supplement: flavocoxid — flavonoid mixture
  Other Names: Limbrel
  Arms: flavocoxid
Drug: Naproxen — non-steroidal anti-inflammatory drug
  Other Names: naprosyn
  Arms: naproxen

SUMMARY:
safety, efficacy and acceptability of Flavocoxid

DETAILED DESCRIPTION:
Safety, Efficacy and acceptability of Flavocoxid (Limbrel) compared with Naproxen in Subjects with Osteoarthritis of the Knee. A Pilot Study

ELIGIBILITY:
Inclusion Criteria:

OA of the knee,K-L grade 2-3 in general good health is currently taking an NSAID or COX-2 inhibitor -

Exclusion Criteria:

pregant or nursing women grade 1 or 4 OA any significant medical condition that in the opinion of the physician might put the subject at risk in this study any form of arthropathy other than OA any condition that might confound the evaluation of the pain, stiffness or function of the target joint intra-articular cotticosteroid inkection in the target joint within 3 month of the screening visit concomitant use of other anti-inflammatory or anti arthritic medication or products(including OTC and herbal preparations) Low dose aspirin for cardio-protection is allowed concomitant use of coumadin or other anticoagulant or anti-platelet medication concomitant use of gastro-protectiv medications including, but not limited to, H2 blockers and proton pump inhibitors, including OTC and herbal products History of allergy to Flavonoids

-

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-03; Primary Completion 2006-07 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
compare efficacy

SECONDARY OUTCOMES:
evaluate safety

CONTACTS AND LOCATIONS:
Overall Officials: Joy Schechtman, DO, Principal Investigator — Sun Valley Arthritis Ltd, 6525 W. Sack Drive Suite 108 Glendale AZ 85308 Phone 623-825-5591 Fax 623; Timothy Truitt, MD, Principal Investigator — MIMA Century Research Associates 65 E. Nasa Blvd. Suite 106 Melbourne FL 32901 Phone 321 723-1203 Fax 321-725-3602
Locations (1):
- Timothy Truitt MD, Melbourne, Florida, United States

REFERENCES:
- [Derived] Levy RM, Saikovsky R, Shmidt E, Khokhlov A, Burnett BP. Flavocoxid is as effective as naproxen for managing the signs and symptoms of osteoarthritis of the knee in humans: a short-term randomized, double-blind pilot study. Nutr Res. 2009 May;29(5):298-304. doi: 10.1016/j.nutres.2009.04.003. PMID 19555810
- See also: Primus Pharmaceuticals, Inc — http://www.primusrx.com